CLINICAL TRIAL: NCT02454634
Title: Targeting IDH1R132H in WHO Grade III-IV IDH1R132H-mutated Gliomas by a Peptide Vaccine - a Phase I Safety, Tolerability and Immunogenicity Multicenter Trial (NOA-16)
Brief Title: Phase I Trial of IDH1 Peptide Vaccine in IDH1R132H-mutated Grade III-IV Gliomas
Acronym: NOA-16
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Tumor Diseases, Heidelberg (Other)
Collaborators: University Hospital Heidelberg (Other); German Cancer Research Center (Other); Neuro-Oncology Working Group of the German Cancer Society (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCT-2013-0216; 2014-000503-27 (EudraCT Number)
Record Dates: First submitted 2015-05-12; First posted 2015-05-27 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2017-09

CONDITIONS: Glioma
Keywords: IDH1R132H; peptide vaccine; immunotherapy; IDH1R132H-mutated glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IDH1 peptide vaccine (Experimental): The IDH1 peptide vaccine is a 20mer peptide encompassing the IDH1R132H-mutated region emulsified in Montanide®. It is injected subcutaneously and administered in combination with topical imiquimod. The vaccine is administered 8 times every 2 or 4 weeks.
  Interventions: Drug: IDH1 peptide vaccine

INTERVENTIONS:
Drug: IDH1 peptide vaccine

SUMMARY:
The NOA-16 trial is the first-in-man trial of the IDH1 (isocitrate dehydrogenase type 1) peptide vaccine targeting the IDH1R132H mutation (amino acid exchange from arginine to glutamine at position 132 of IDH1). The aim of this trial is to evaluate the safety and tolerability of and immune response to the IDH1 peptide vaccine in patients with IDH1R132H-mutated, WHO grade III-IV gliomas.

DETAILED DESCRIPTION:
The patient population will be molecularly defined and include IDH1R132H mutant grade III and IV gliomas without co-deletion of 1p/19q and with loss of alpha-thalassemia/mental retardation syndrome X-linked (ATRX) expression.

Within this trial, the IDH1 peptide vaccine will be administered to 39 patients.

In treatment group 1 vaccination treatment will be done alone starting 4-6 weeks post radiotherapy. In treatment groups 2 and 3 vaccination treatment will be done in parallel with temozolomide (TMZ) chemotherapy starting at day 10 of the 4th TMZ cycle (treatment group 2) or at day 10 of the 1st TMZ cycle post concomitant radiochemotherapy (treatment group 3).

ELIGIBILITY:
Inclusion Criteria:

* Patients present with histologically confirmed diagnosis of an IDH1R132H-mutated glioma (with or without measurable residual tumor after tumor resection or biopsy)
* Histology may be astrocytoma, oligodendroglioma, or oligoastrocytoma WHO grade III or IV
* Absence of chromosomal 1p/19q co-deletion in the tumor tissue
* Loss of nuclear ATRX expression in the tumor tissue (partial loss allowed)
* Availability of tumor tissue for molecular screening (FFPE bulk tissue or biopsy)
* Patients have received radiotherapy (54 - 60 Gy) alone, 3 cycles of chemotherapy with TMZ (150-200 mg/m2, 5/28 days) or standard combined radiochemotherapy with TMZ prior to enrollment.
* Patients should be immunocompetent (i.e. no concomitant treatment with dexamethasone (or equivalent), or receive stable/decreasing steroid levels not exceeding 2 mg/day dexamethasone (or equivalent) during the last 3 days prior to clinical screening; no severe lymphopenia)
* ≥18 years old, smoking or non-smoking, of any ethnic origin and gender
* Karnofsky Performance Status ≥ 70
* Ability of patient to understand character and individual consequences of the clinical trial
* Evidence of two informed consent documents personally signed and dated by the patient (or a witness in case the patient is unable to write) covering the molecular screening procedure (short IC) and the remaining trial-related procedures (extended IC) and indicating that the patient has been informed of all pertinent aspects of the study and that the patient consents to participate in the trial.
* Women of child-bearing potential (WOCBP; i.e., those who have not undergone a hysterectomy, bilateral salpingectomy and bilateral oophorectomy or who have not been post-menopausal for at least 24 consecutive months) must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of the investigational medicinal product (IMP).
* WOCBP must be using an effective method of birth control to avoid pregnancy throughout the study and for 24 weeks after the last dose of the IMP. This includes two different forms of effective contraception (e.g., hormonal contraceptive and condom, IUD/IUS and condom) or sterilization, resulting in a failure rate less than 1% per year.
* Men must be willing and able to use an effective method of birth control throughout the study for up to 24 weeks after the last dose of the IMP, if their sexual partners are WOCBP (acceptable methods see above).
* Patients who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* Progressive (incl. pseudoprogression) or recurrent disease after radiation therapy, chemotherapy or radiochemotherapy based on local MRI assessment
* Previous or concurrent experimental treatment for the tumor. This includes local therapies such as interstitial radiotherapy or local chemotherapy (i.e. BCNU wafers), loco-regional hyperthermia, and antiangiogenic therapy (such as bevacizumab)
* Antitumor treatment other than standard radiotherapy and/or standard TMZ chemotherapy. Daily metronomic TMZ or intensified dosing scheduled as a substitute for maintenance TMZ cycles are not allowed. (Dose reductions of standard TMZ chemotherapy are allowed.)
* Abnormal (≥ Grade 2 CTCAE v4.0) laboratory values for hematology, liver and renal function (serum creatinine). In detail the following values apply as exclusion criteria:

  1. Hemoglobin < 10 g/dL (6.2 mmol/L)
  2. White blood cell count (WBC) decrease (<3.0 x 109/L) or increase (>10.0 x 109/L)
  3. Absolute neutrophil count (ANC) decrease (< 1.5 x 109/L)
  4. Platelet count decrease (< 75 x 109/L)
  5. Bilirubin > 1.5 x ULN (upper limit of normal according to the performing lab's reference range)
  6. ALT > 3 x ULN
  7. AST > 3 x ULN
  8. GGT > 2.5 x ULN
  9. Serum creatinine increase (> 1.5 x ULN)
* Pregnancy and lactation
* Patients with history or presence of HIV and/or HBV/HCV
* Patients with history or known presence of tuberculosis
* Patients with severe infection(s) or signs/symptoms of infection within 2 weeks prior to the first administration of the study drug
* Patients who have received a live, attenuated vaccine within 4 weeks prior to the first administration of the study drug
* Patients with a prior solid organ transplantation or haematopoietic stem cell transplantation
* History of hypersensitivity to the IMP or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the IMP
* Participation in other clinical trials or their observation period during the last 30 days before the first administration of the IMP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-09-19 (Actual); Study Completion 2017-09-19 (Actual)

PRIMARY OUTCOMES:
safety and tolerability of repeated fixed dose vaccinations of the IDH1 peptide vaccine administered with topical imiquimod (Aldara®) assessed by Regime Limiting Toxicity (RLT). | 15 months
  Primary safety endpoint is the Regime Limiting Toxicity (RLT).
immunogenicity of the IDH1 peptide vaccine | 15 months
  The primary immunogenicity endpoint is the presence of an IDH1R132H-specific T-cell and/or antibody response at any time point during the trial measured by IFN-gamma ELISpot and ELISA, respectively (response Yes/No).

SECONDARY OUTCOMES:
immunogenicity by assessing the IDH1R132H-specific T-cell and antibody response | 15 months
progression-free survival (PFS) | 15 months
overall response rate (ORR) | 15 months
association between immunogenicity (IDH1R132H-specific T-cell and antibody response) and the clinical outcome parameters (ORR, PFS) | 15 months
  assessed by Logistic regression and Proportional Hazard models

CONTACTS AND LOCATIONS:
Overall Officials: Michael Platten, MD, Principal Investigator — University Hospital Heidelberg, Neurology Clinic; Neurooncology Program at the NCT
Locations (8):
- Germany (8):
  - Charité Berlin, Neurosurgery, Berlin
  - University Hospital Dresden, Neurosurgery, Dresden
  - University Hospital Essen, Internal Medicine, Essen
  - University Hospital Frankfurt, Neurooncology, Frankfurt am Main
  - University Hospital Freiburg, Neurosurgery, Freiburg im Breisgau
  - University Hospital Heidelberg, Neurology Clinic, Heidelberg
  - LMU, University Hospital Munich, Munich
  - University Hospital Tuebingen, Neurooncology, Tübingen

REFERENCES:
- [Derived] Platten M, Bunse L, Wick A, Bunse T, Le Cornet L, Harting I, Sahm F, Sanghvi K, Tan CL, Poschke I, Green E, Justesen S, Behrens GA, Breckwoldt MO, Freitag A, Rother LM, Schmitt A, Schnell O, Hense J, Misch M, Krex D, Stevanovic S, Tabatabai G, Steinbach JP, Bendszus M, von Deimling A, Schmitt M, Wick W. A vaccine targeting mutant IDH1 in newly diagnosed glioma. Nature. 2021 Apr;592(7854):463-468. doi: 10.1038/s41586-021-03363-z. Epub 2021 Mar 24. PMID 33762734